CLINICAL TRIAL: NCT05413252
Title: Facilitation of Team-based Care to Improve HTN Management and Outcomes
Brief Title: Team-based Care to Improve Hypertension
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: New York City Department of Health and Mental Hygiene (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-FY2022-6555
Record Dates: First submitted 2022-06-03; First posted 2022-06-09 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: team-based care; practice facilitation; implementation
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The study is conducting a stepped-wedge design RCT trial. Practices will be randomized into the study into one of three waves.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Current Practice (No Intervention): Practices will deliver care as usual and patients at these sites receive standard HTN care delivered.
- Practice Facilitation (Active Comparator): Practices review coaching and support from a trained practice facilitator. This includes 24 site visits in which facilitators meet with staff to work on implementing system changes to improve hypertension management.
  Interventions: Other: Practice Facilitation

INTERVENTIONS:
Other: Practice Facilitation — Practices will be assigned a practice facilitator who will support practices in implementing all practice redesign components associated with TBC for HTN management.
  Other Names: team-based care implementation
  Arms: Practice Facilitation

SUMMARY:
The study is a stepped-wedge cluster randomized control trial to compare the effect of Practice Facilitation in 90 small-to-medium sized independent primary care practices on the adoption of team-based care.

DETAILED DESCRIPTION:
The study is designed to transform health care delivery by helping smaller independent practices to adopt team-based care. The study will use a stepped-wedge cluster randomized control trial to compare the effect of Practice Facilitation in small-to-medium sized independent primary care practices on the adoption of team-based care aimed at improving hypertension management and blood pressure control. The study will recruit approximately 90 practices which receive practice facilitation to support the adoption of team-based care. Sites are then randomly assigned to one of three waves in which they cross over to the intervention phase. Waves are separated by 6 months and the intervention period lasts 12 months. This is followed by a phase in which sustainability of TBC and BP control is assessed. Each practice will be assigned a practice facilitator and will be required to identify a site champion who will be a member of the team. PF activities will support practices in implementing all practice redesign components associated with TBC for HTN management through training, coaching, modeling TBC, and making changes to systems where necessary to support TBC. Data collection for the primary outcome (adoption of TBC) occurs immediately prior to the beginning of the next 6-month wave. BP outcome data is collected over the 6-month period prior to the next wave. Outcomes will be measured every 6 months in all clusters at every time period so that each cluster provides data points in both the control and intervention conditions.

ELIGIBILITY:
Inclusion Criteria:

* One to 5 healthcare providers
* Minimum of 2 non-physician staff available at any time
* Use an electronic health record (EHR) system to deliver care
* Have no plans to participate in another CVD-related quality improvement initiative during the study
* Willing to identify a "physician champion" or staff member to collaborate on all aspects of the intervention
* Have a minimum of 200 patients on their practice panels that have hypertension that are managed by the practice
* Agree to study terms including randomization, data sharing, participation in PF, and completion of surveys

Exclusion Criteria:

* Five or more healthcare providers
* Do not have sufficient non-physician staff on board to adopt team-based care
* Do not use an electronic health record (EHR) system to deliver care
* Participation or planned participation in another CVD-related improvement initiative during the time of the study
* Unwilling to identify a "physician champion" or staff member to collaborate on all aspects of the intervention
* Less than 200 patients on their practice panel that have hypertension that are managed by the practice.
* Failure to agree to study terms including randomization, data sharing, participation in PF, and completion of surveys
* Primary care practices which are unable to provide patient level BP data for 6 months prior to enrolling into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of practices that adopt team-based care as assessed by the Primary Care Team Dynamic Survey and Team Process - Monitoring Progress Toward Goals sub-scale. | 12 months
  Five core constructs of team-based care will be measured (clear roles, communication, mutual support, measurable processes and outcomes, and shared goals) by Primary Care Team Dynamic Survey and Team Process - Monitoring Progress Toward Goals sub-scale.

SECONDARY OUTCOMES:
Percentage of with a diagnosis of hypertension who have a BP <140/90 (JNC Guidelines) as assessed through EHRs reports. | 12 months
  Percentage of patients 18 - 85 years of age who had a diagnosis of hypertension prior to and overlapping the measurement period and whose most recent blood pressure was adequately controlled (< 140/90 mmHg) during the measurement period.

CONTACTS AND LOCATIONS:
Overall Officials: Donna Shelley, MD, Principal Investigator — NYU School of Global Public Health
Locations (2):
- United States (2):
  - New York University, New York, New York
  - New York University School of Global Public Health, New York, New York

REFERENCES:
- [Result] Shelley DR, Brown D, Cleland CM, Pham-Singer H, Zein D, Chang JE, Wu WY. Facilitation of team-based care to improve HTN management and outcomes: a protocol for a randomized stepped wedge trial. BMC Health Serv Res. 2023 May 31;23(1):560. doi: 10.1186/s12913-023-09533-1. PMID 37259081